CLINICAL TRIAL: NCT01334788
Title: Sleep Deprivation and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, MD, PhD, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-006780; R21HL096071-02 (NIH)
Record Dates: First submitted 2010-10-26; First posted 2011-04-13 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation; sleep restriction
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleep deprivation (Experimental): These are subjects who are randomized to undergo sleep deprivation.
  Interventions: Other: sleep deprivation
- Normal sleep (Other): These are subjects who are randomized to sleep normally.
  Interventions: Other: Normal sleep

INTERVENTIONS:
Other: sleep deprivation — Sleep restriction
  Other Names: sleep restriction
  Arms: sleep deprivation
Other: Normal sleep — These are subjects who are randomized to sleep normally.
  Other Names: control
  Arms: Normal sleep

SUMMARY:
Chronic sleep deprivation may constitute an important and potentially correctable behavioral factor in the alarming increase in obesity. There are no definitive experimental studies in humans showing whether sleep deprivation indeed contributes to increased energy intake and/or reduced energy expenditure. The investigators propose a series of novel studies to investigate abnormalities in energy homeostasis imparted by sleep deprivation. The investigators will measure food intake, energy expenditure (basal metabolic rate, thermal effect of food, and non-exercise activity thermogenesis), and neurohormone levels in 24 healthy subjects with normal BMI (20-25 kg/m2). Twelve subjects (6 men and 6 women) will be randomized to sleep deprivation. Measurements will be compared to those obtained in 12 subjects who are randomized to a control group, and are not sleep deprived. The investigators will test the following hypotheses: 1. That sleep deprivation results in positive energy balance (increased caloric intake and decreased energy expenditure, as reflected by decreased non-exercise activity thermogenesis). 2. That dysregulation of appetite and energy expenditure is associated with changes in molecules controlling appetite and metabolism. 3. That changes associated with 8 days of modest sleep deprivation resolve, at least in part, over a 4 day recovery period.

DETAILED DESCRIPTION:
The demands of present day living have placed a high premium on time. Voluntary sleep curtailment is endemic and many adults typically sleep an average of six hours per night. Observational data suggest that short sleep duration is associated with a greater likelihood of being obese. Low grade chronic sleep deprivation may constitute an important and potentially correctable behavioral factor in the alarming increase in obesity. There are no definitive experimental studies in humans showing whether sleep deprivation indeed contributes to increased energy intake and/or reduced energy expenditure. The investigators propose a series of novel studies to investigate abnormalities in energy homeostasis imparted by sleep deprivation. These studies combine state-of-the-art techniques for monitoring sleep, food intake, energy expenditure and neuroendocrine energy regulation. The investigators will measure food intake, energy expenditure (basal metabolic rate, thermal effect of food, and non-exercise activity thermogenesis), and neurohormone levels in 24 healthy subjects with normal BMI (20-25 kg/m2). Twelve subjects (6 men and 6 women) will be randomized to sleep deprivation. After a 3 day baseline evaluation, these subjects will undergo 8 days of modest sleep deprivation followed by a 4 day recovery period. Measurements will be compared to those obtained in 12 subjects who are randomized to a control group, and are not sleep deprived. Sleep deprived and control subjects will be comparable for age and gender and will undergo similar monitoring and measurements in the Clinical Research Unit over the same duration. The investigators will test the following hypotheses: 1. That sleep deprivation results in positive energy balance (increased caloric intake and decreased energy expenditure, as reflected by decreased non-exercise activity thermogenesis). 2. That dysregulation of appetite and energy expenditure is associated with changes in molecules controlling appetite and metabolism. 3. That changes associated with 8 days of modest sleep deprivation resolve, at least in part, over a 4 day recovery period. This exploratory application builds on established research programs addressing first, neuroendocrine mechanisms in sleep and obesity, and second, the regulation of energy intake and energy expenditure in humans. These studies will provide novel and important insights into whether sleep deprivation promotes increased food intake and/or reduced activity levels, and into the potential role of molecules that regulate appetite and metabolism. PUBLIC HEALTH RELEVANCE: The investigators propose to examine whether two weeks of modest sleep restriction results in increased food intake and decreased energy expenditure, thus potentially predisposing to obesity. These findings will help explain whether the reduced sleep duration in the general population may be contributing to the current epidemic of obesity, and suggest novel strategies for weight control.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be sedentary. Sedentary will be defined as those with an occupational calorie expenditure that is not estimated at greater than 50% above basal (desk job or light activity at work: on feet 30-50% of the work day) and whose exercise activity is defined as sedentary according to a self-reported activity questionnaire, and confirmed by actigraphy measurements. Sedentary lifestyle will be defined as fewer than four 20 min episodes of moderate or vigorous intensity activity in the previous four weeks.

Exclusion Criteria:

* We will exclude subjects who have any medical or psychiatric disorders, including history of anxiety or depression, and those taking any medications.
* Those found to have depression on a depression screening tool (BDI-II) will be excluded.
* Current smokers will be excluded.
* All female subjects will undergoing a screening pregnancy test and excluded if positive.
* Subjects found to have significant sleep disorders will be excluded. -
* Subjects found to have occult coronary artery disease by exercise treadmill testing will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sleep Deprivation results in positive energy balance | 15 days
  The investigators are testing the hypothesis that sleep deprivation results in increased caloric intake (calories from food consumed) and reduced energy expenditure (calories burned), resulting in a net positive energy balance.

CONTACTS AND LOCATIONS:
Overall Officials: Erik K St Louis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Calvin AD, Covassin N, Kremers WK, Adachi T, Macedo P, Albuquerque FN, Bukartyk J, Davison DE, Levine JA, Singh P, Wang S, Somers VK. Experimental sleep restriction causes endothelial dysfunction in healthy humans. J Am Heart Assoc. 2014 Nov 25;3(6):e001143. doi: 10.1161/JAHA.114.001143. PMID 25424573
- [Derived] Calvin AD, Carter RE, Adachi T, Macedo PG, Albuquerque FN, van der Walt C, Bukartyk J, Davison DE, Levine JA, Somers VK. Effects of experimental sleep restriction on caloric intake and activity energy expenditure. Chest. 2013 Jul;144(1):79-86. doi: 10.1378/chest.12-2829. PMID 23392199